CLINICAL TRIAL: NCT07378332
Title: Towards Causal Mapping of Episodic Memory iEEG Networks Via Multi-method Brain Stimulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Northwestern University, Chicago, IL (Unknown); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB24-0486
Record Dates: First submitted 2026-01-16; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Memory Performance; Hippocampal Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TMS stimulation using HITS (Experimental): Hippocampal indirectly targeted stimulation (HITS) will be applied in patients with epilepsy undergoing intracranial electroencephalography (iEEG) monitoring. iEEG signals of episodic memory behavioral performance will be obtained from clinical macroelectrodes and research microelectrodes in a specialized memory task involving encoding and retrieval of naturalistic scenes along with eye-movement tracking. Memory behaviors of interest will include recollection during old/new decisions and spatiotemporal replay of eye-movement patterns. HITS will be applied for ~2 s immediately before each scene onset during encoding, using parameters that have yielded enhanced versus impaired performance in this experiment design
  Interventions: Other: TMS electrical stimulation parameters during cognitive and memory demands
- DES stimulation using HITS parameters (Experimental): We will test the behavioral significance of iEEG correlates of memory enhancement and impairment using a rigorous approach involving DES. Direct electrical stimulation (DES) parameters will be identified that reproduce as closely as possible the iEEG signatures of memory enhancement or impairment caused by HITS. This will be accomplished using a closed-loop machine learning approach to maximize the similarity of the iEEG signals evoked by DES and the iEEG signals evoked by HITS, during memory encoding.
  Interventions: Other: DES electrical stimulation parameters during cognitive and memory demands
- Normative model of DES (Experimental): We will develop, test, and refine for future experiments a normative model of DES parameters to achieve experimental bi-directional manipulation of iEEG correlates of episodic memory. We will identify common features of the DES parameters that were algorithmically determined to mimic the iEEG signals of memory enhancement or impairment by HITS in the Experiment 2 dataset. Analyses will account for individual differences in stimulated electrode locations, in iEEG functional connectivity of stimulated electrodes, in the success of behavioral modification, and in the accuracy of mimicking the iEEG effects of HITS, to enable predictions about how to apply DES parameters in stimulation-naïve subjects given their idiosyncratic electrode placements and brain activity patterns.
  Interventions: Other: DES electrical stimulation parameters during cognitive and memory demands

INTERVENTIONS:
Other: TMS electrical stimulation parameters during cognitive and memory demands — Study conditions will involve electrical stimulation delivered through non-invasive TMS. These different stimulation parameters will include the presence of stimulation (no stimulation versus stimulation) and the location of stimulation.
  Arms: TMS stimulation using HITS
Other: DES electrical stimulation parameters during cognitive and memory demands — Study conditions will involve direct electrical stimulation delivered through implanted iEEG electrodes. These different stimulation parameters will include the presence of stimulation (no stimulation versus stimulation) and the location of stimulation across the same electrode or a different electrode.
  Arms: DES stimulation using HITS parameters; Normative model of DES

SUMMARY:
Human intracranial electroencephalography (EEG) can provide brain-activity correlates of memory with high spatial and temporal resolution. This project will test functional relevance of these neural signals for memory behavioral performance using novel noninvasive and invasive stimulation methods. Findings will advance understanding of brain mechanisms for memory, as is needed to accelerate progress in the treatment of memory disorders.

DETAILED DESCRIPTION:
Episodic memory impairment occurs when diseases impact the hippocampus and its network of interacting brain areas. Better understanding of brain mechanisms for memory is required to development treatments. This project will develop experimental approaches that use stimulation to manipulate brain-behavior relationships in humans and thereby directly test how the hippocampal network supports memory. Intracranial electroencephalography (iEEG) provides opportunities to study the neural basis of memory with high spatial and temporal resolution. Many experiments have identified iEEG signals associated with memory, for instance by comparing instances of memory success to failure. However, the functional relevance of these signals remains unclear, as such comparisons can identify signals of extraneous, co-occurring, cognitive processes. A routine approach to address this limitation in the behavioral neurosciences is via bi-directional manipulations, i.e., exogenous enhancement or inhibition of the putative neural process and tests of corresponding enhancement or inhibition of behavioral performance. This approach has been underutilized in human iEEG memory research, in part due to difficulties in reliably influencing memory or neural signals given currently available manipulations, such as direct electrical stimulation (DES) through iEEG electrodes. As a route to achieve bi-directional manipulation experiments in human iEEG memory research, this project utilizes a noninvasive electromagnetic stimulation tool that reliably and robustly influences hippocampal network activity and memory performance, called "hippocampal indirectly targeted stimulation" (HITS). HITS will be used with iEEG for the first time to identify activity patterns of the hippocampal network related to memory behavioral performance enhancement versus impairment. To rigorously test for behavioral relevance, we will use a closed-loop machine-learning approach to identify DES parameters that reproduce the hippocampal-network iEEG activity patterns generated by HITS, and then test whether delivery of DES to enhance or inhibit these hippocampal-network iEEG activity patterns produces corresponding enhancement versus impairment of memory behavioral performance. Thus, bidirectional manipulation will be used to directly/causally test iEEG signals of memory behavior. Group-level modeling of DES parameters that mimic the effects of HITS will be used to broaden the accessibility of bidirectional manipulations for future research that tests memory mechanisms in larger iEEG samples across multiple sites that lack the technical capability for HITS. Across three sites, will test whether bi-directional manipulations of hippocampal-network activity involvement in memory performance are more successful for HITS-informed DES versus DES based on a priori hypotheses. This exploratory project will thus build a foundation for future studies to rigorously test hippocampal-network support of memory behavioral performance using bi-directional experimental manipulations and will establish a collaboration of multidisciplinary researchers across multiple institutions to perform this innovative mechanistic memory research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years old
* Native English speakers
* Normal or corrected-to-normal near and far vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Power of theta-band hippocampal iEEG activity | Measured during the performance of the task while research activities are completed. Measurement will take 2 to 4 hours on a single day
  iEEG is used to measure local brain electrical activity evoked by task conditions. We will record and analyze the power of theta-band hippocampal iEEG activity
iEEG activity between hippocampus and the stimulated electrode | Measured during the performance of the task while research activities are completed. Measurement will take 2 to 4 hours on a single day
  iEEG is used to measure local brain electrical activity evoked by task conditions. We will record and analyze the synchrony of iEEG activity between hippocampus and the stimulated electrode.
Memory task performance | The memory task is administered before, during and/or after stimulation from transcranial magnetic stimulation (TMS) or direct electrical stimulation (DES). The memory task will take 2 to 4 hours in a single day.
  Subjects attempt to discriminate studied from novel (foil) scenes and object images

CONTACTS AND LOCATIONS:
Overall Officials: Joel Voss, PhD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No